CLINICAL TRIAL: NCT05662527
Title: Efficacy of Immunotherapy in Patients With MMR-deficient Localized Colon Cancer Scheduled for Curative Surgery - A Prospective, Phase II Study
Brief Title: Response to Immunotherapy in MMR-deficient Localized Colon Cancer
Acronym: RESET-C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Camilla Qvortrup (Other)
Collaborators: Zealand University Hospital (Other); Odense University Hospital (Other); Vejle Hospital (Other); Herlev and Gentofte Hospital (Other); Bispebjerg Hospital (Other); Aalborg University Hospital (Other); Horsens Hospital (Other); Randers Regional Hospital (Other); Aarhus University Hospital (Other)
Responsible Party: Sponsor-Investigator, Camilla Qvortrup, Senior physician oncology, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 011121
Record Dates: First submitted 2022-11-24; First posted 2022-12-22 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Colon Cancer
Keywords: Localized colon cancer; dMMR; Immunotherapy; Biomarkers
MeSH Terms: conditions — Colonic Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant pembrolizumab (Experimental): Pembrolizumab
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — One dosage of 4mg/kg (maximum of 400mg)
  Other Names: Keytruda

SUMMARY:
The aim of this study is to evaluate the safety and efficacy of neoadjuvant treatment with pembrolizumab before colonic resection in patients with early-stage (I-III) deficient mismatch repair (dMMR) colon cancer (CC).

DETAILED DESCRIPTION:
The trial is designed as an investigator-initiated, multicenter, prospective, single arm phase II study in patients with stage I-III dMMR CC scheduled for intended curative surgery to determine the efficacy of immunotherapy using pembrolizumab in the neoadjuvant setting. Patients will receive one dose of pembrolizumab (dosage of 4mg/kg, maximum of 400mg) following diagnosis. After 3 weeks a re-evaluation (to assess tumor response) will be performed, followed by standard surgery for resection of the tumor. Surgery will therefore be performed within 3 to 5 weeks after the dose of pembrolizumab treatment. Following the surgical resection the patients may receive post-operative chemotherapy in accordance with the clinical decision. The patients will be followed as per the standard Danish guidelines with CT scans at 1 and 3 years after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed localized dMMR stage cT1N0M0 to cT4N2M0 (stage I to III) colon carcinoma.
2. Indication for elective curative intended surgery without neoadjuvant chemotherapy.
3. Age of ≥ 18 years.
4. Written informed consent.
5. Eastern Cooperative Oncology Group performance status of 0 or 1.
6. Adequate bone marrow function defined as:

   * Hemoglobin ≥ 6.2 mmol/L or ≥ 10 g/dL.
   * Absolute neutrophil count ≥ 1.5 × 109/L.
   * Platelet count ≥ 100 × 109/L.
7. Adequate kidney function defined as:

   o Estimated glomerular filtration rate ≥ 60 mL/min or creatinine ≤1.5 × upper limit of normal (ULN).
8. Adequate liver function defined as:

   * Total bilirubin: ≤ 1.5 × ULN.
   * Alanine aminotransferase: ≤ 2.5 × ULN.
   * Alkaline phosphatase: ≤ 2.5 × ULN.
9. Follow the conditions regarding fertility, pregnancy, and lactation:

   * Female and male participants of reproductive potential (PORP) must agree to avoid becoming pregnant or impregnating a partner, respectively, while receiving pembrolizumab and for 120 days after the dose.
   * PORPs must use, or have their partner use, an acceptable method of contraception e.g. intrauterine device, contraceptive rod implanted into the skin, or hormonal contraceptive and male condom during heterosexual activity, while receiving pembrolizumab and for 120 days after the dose.
   * Women of reproductive potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L HCG) within 72 hours prior to receiving pembrolizumab.
   * Women must not be breastfeeding.

Exclusion Criteria:

1. Any serious or uncontrolled medical disorder that, in the opinion of the investigator or treating physician, may increase the risk associated with study participation, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results.
2. Autoimmune disorders (except thyroiditis with replacement therapy and type I diabetes mellitus).
3. Prior treatment with ICIs or any other antibody/drug specifically targeting the T-cell co-stimulation or checkpoint pathways.
4. A known history of Human Immunodeficiency Virus, active chronic, or acute Hepatitis B or Hepatitis C.
5. A condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
6. Prior participation in another trial with an investigational medicinal product.
7. Received live vaccines within 30 days prior to pembrolizumab trial treatment. Seasonal influenza vaccines for injection are allowed.
8. A history of allergy to study drug components or a history of severe hypersensitivity reaction to any monoclonal antibody.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2023-02-22 (Actual); Primary Completion 2024-06-06 (Actual); Study Completion 2024-06-06 (Actual)

PRIMARY OUTCOMES:
Pathological complete response (pCR) | Tumour specimen evaluated within 2 weeks after surgery.
  Number of patients with pCR evaluated according to the Mandard tumour regression grading system

SECONDARY OUTCOMES:
Safety and tolerability of pembrolizumab administered before surgery | Up to approximately 9 weeks
  Determined by the incidence and severity of treatment related adverse events according to CTCAE version 5.0
Postoperative surgical complications | Before and up to 4 weeks after surgery
  Number and severity of postoperative surgical complications determined by Clavien-Dindo classification system.
Immunohistochemistry analysis of markers including CD3, CD8, and PD-L1 | Baseline compared to the surgical specimen at 3-5 weeks
  Assessment of potential predictive biomarker by investigating immunological markers across pre- and post-treatment biopsies and sequential blood samples.
Methylated circulating cell-free DNA | Up to approximately 9 weeks
  Treatment response evaluated by methylated circulating cell-free DNA (cfDNA) specific for CC analysed across sequential blood samples using the TriMeth test
Gene expression by mRNA | Baseline compared to the surgical specimen at 3-5 weeks
  To quantify the expression of genes central to the tumour microenvironment and immune evasion of cancer among others

OTHER OUTCOMES:
TCR sequencing | Baseline compared to 3-5 weeks after pembrolizumab and 2-3 weeks after surgery
  To investigate the role of the adaptive immune system in mediating the effect of pembrolizumabrepertoire, CT-scans, endoscopic photo documentation, and patient journals will be analysed with the purpose of identifying biomarkers for predicting pCR.
CT chest/abdomen scans | 1-5 weeks before pembrolizumab and 3-5 weeks after pembrolizumab
  Evaluated by a multidisciplinary team and centralized comity of radiologists according to the RECIST 1.1 criteria as well as cTNM staging
Endoscopic tumour assessment | 1-5 weeks before pembrolizumab and 3-5 weeks after pembrolizumab
  Assessed by a systematic approach including the Paris and NICE classifications

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Qvortrup, MD, PhD, Study Director — Rigshospitalet, Denmark; Ismail Gögenur, Professor, Principal Investigator — Zealand University Hospital
Locations (1):
- Zealand University Hospital, Roskilde, Denmark

IPD SHARING:
Plan to Share IPD: Yes
In accordance with good academic practice, the study data (health data and genomic data) is planned to be transferred in anonymized form to the secure database European Genome-Phenome Archive (EGA). This will happen after the study has been completed. The purpose is to enable sharing of the data with other research groups for future research, inside and outside of Denmark. In all cases, data access decisions will be made by the study protocol committee. Data sharing will be conducted in accordance with the European data protection regulations, including The Danish Data Protection Act and the General Data Protection Regulation. The EGA is part of the European ELIXIR research infrastructure, which is partly funded by the European Commission.
Supporting Information: Study Protocol, ICF
Time Frame: Planned to begin approximately 6 months end ending approximately 5 years after publication of the final article.
Access Criteria: Reasonable request. In all cases, data access decisions will be made by the study protocol committee.

REFERENCES:
- [Derived] Gogenur I, Justesen TF, Tarpgaard LS, Bulut M, Hansen TF, Jensen LH, Rahr HB, Kirkegaard T, Balsevicius L, Raskov H, Petersen PC, Eriksen JR, Salomon S, Fiehn AK, Brandsborg S, Gotschalck KA, Emmertsen KJ, Born PW, Thorlacius-Ussing O, Lauritzen MB, Olesen RK, Poulsen LO, Lykke J, Schou J, Buskov L, Krarup PM, Andersen CL, Pfeiffer P, Qvortrup C. Neoadjuvant Pembrolizumab in Stage I-III Deficient Mismatch Repair Colon Cancer: A Clinical Trial. Ann Surg. 2024 Dec 18. doi: 10.1097/SLA.0000000000006611. Online ahead of print. PMID 39692004
- [Derived] Justesen TF, Gogenur I, Tarpgaard LS, Pfeiffer P, Qvortrup C. Evaluating the efficacy and safety of neoadjuvant pembrolizumab in patients with stage I-III MMR-deficient colon cancer: a national, multicentre, prospective, single-arm, phase II study protocol. BMJ Open. 2023 Jun 22;13(6):e073372. doi: 10.1136/bmjopen-2023-073372. PMID 37349100